CLINICAL TRIAL: NCT04376242
Title: The Utilization of Virtual Reality Technology Versus Standard of Care During Pediatric Oral Food Challenge: a Pilot Study
Brief Title: Virtual Reality Technology Versus Standard Technology During Pediatric Oral Food Challenge
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Resources not available to continue study
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sayantani B. Sindher, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 56108
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Food Allergy in Children; Food Allergy
Keywords: food allergy; oral food challenge; virtual reality
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality then standard technology (Experimental): patients randomized to this arm will first use virtual reality (VR) during and oral food challenge and then use standard technology during a second oral food challenge
  Interventions: Behavioral: use of virtual reality; Behavioral: use of standard technology
- standard technology then virtual reality (Active Comparator): patients randomized to this arm will first use standard technology during and oral food challenge and then use virtual reality during a second oral food challenge
  Interventions: Behavioral: use of virtual reality; Behavioral: use of standard technology

INTERVENTIONS:
Behavioral: use of virtual reality — The intervention is a virtual reality program designed to immerse participants in a gaming experience to improve anxiety and fear during an oral food challenge.
Behavioral: use of standard technology — the active comparator group will be allowed standard technology for distraction during oral food challenge which can include TV, non-VR gaming, tablets and smart phones.

SUMMARY:
The purpose of this study is to determine if non-invasive distracting devices (Virtual Reality headset) are more effective than the standard of care of utilizing existing technologies that are currently more common in food allergy research treatment and clinics (i.e. television and patients' personal electronic devices) for decreasing levels anxiety and fear in pediatric patients undergoing oral food challenge (OFC) and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 5 and 17
* Willing to participate in both the VR and standard of care technology conditions
* Able to consent or have parental consent
* Undergoing at least two Oral Food Challenges within the window of recruitment at the Sean N. Parker Center

Exclusion Criteria:

* People who do not consent
* Significant Cognitive Impairment
* History of Severe Motion Sickness
* Current Nausea
* Seizures
* Visual Problems
* Non-English Speaking
* Patients who clinically unstable or requires urgent/emergent intervention
* ASA class 4 or higher

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Children's Fear Scale Score Before and After OFC dosing | measurements occur at single time points before and after each food challenge with approximately 4-6 hours between measurements. Thus 4 discrete measurements will be taken over two food challenges which will occur approximately one week apart.
  The Children's Fear Scale (CFS) is used to measure the anxiety or fear level of the children. The one-item scale consists of a row of five sex neutral faces ranging from a no fear (neutral) face on the far left to a face showing extreme fear on the far right.
Change in Childhood Anxiety Meter Score Before and After OFC dosing | Before and after each evaluation (approximately 4-6 hours between measurements at each visit, with visits approximately 1 week apart)
  The Childhood Anxiety Meter brief measure of the current level of anxiety in a child using a visual scale (thermometer that is colored to the level anxiety, higher thermometer level means more anxiety).

SECONDARY OUTCOMES:
Level of Immersion after OFC | After each evaluation (approximately 1 week apart)
  Modified scale to assess cognitive absorption as a measure of immersion in the technology.
Level of satisfaction - participant, caregiver and provider | After each evaluation (approximately 1 week apart)
  Patient, caregiver and provider satisfaction after dosing will be assessed through a custom satisfaction evaluation form, with categorical responses to questions tailored to specific challenges during OFC such as the time it takes to administer a dose, how well a patient complies with dosing, and how available technology may influence patient and caregiver desire to continue with a study.

CONTACTS AND LOCATIONS:
Overall Officials: Sayantani Sindher, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share.